CLINICAL TRIAL: NCT02327312
Title: Multicenter Investigation of Trabecular Micro-Bypass Stents vs. Laser Trabeculoplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC-004
Record Dates: First submitted 2014-11-06; First posted 2014-12-30 (Estimated); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Primary Open-Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Stents; Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical (Experimental): Implantation of two Trabecular Meshwork stents into the study eye
  Interventions: Device: Stents
- Laser (Active Comparator): Laser Trabeculoplasty
  Interventions: Procedure: Laser; Device: Laser Trabeculoplasty

INTERVENTIONS:
Device: Stents — Two Trabecular meshwork Micro-Bypass stents into the study eye
  Arms: Surgical
Procedure: Laser — Laser Trabeculoplasty
  Arms: Laser
Device: Laser Trabeculoplasty
  Arms: Laser

SUMMARY:
To evaluate the safety and effectiveness of Trabecular Micro-Bypass stents (two stents per study eye) vs. laser trabeculoplasty, in subjects with open angle glaucoma

ELIGIBILITY:
Inclusion Criteria:

* Open angle Glaucoma

Exclusion Criteria:

* Active corneal inflammation or edema
* Choroidal detachment, effusion, choroiditis

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
IOP reduction | up to 24 months

SECONDARY OUTCOMES:
% IOP reduction | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Stephens, OD, Study Chair — Glaukos Corporation
Locations (9):
- United States (9):
  - Glendale, Arizona
  - Fayetteville, Arkansas
  - Hemet, California
  - Cape Coral, Florida
  - Elizabeth City, North Carolina
  - Memphis, Tennessee
  - Fort Worth, Texas
  - San Antonio, Texas
  - Racine, Wisconsin

REFERENCES:
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114